CLINICAL TRIAL: NCT06777355
Title: Liver Infusion Flow Evaluation With ultraSound for Assessment of Right Ventricular Function: a Single cEnter Cohort Study (LIFESAVE)
Brief Title: Association Between Portal Flow Pulsatility and Right Ventricular Dysfunction in the Postoperative Period of Cardiac Surgery
Acronym: LIFESAVE
Status: Completed | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/04
Record Dates: First submitted 2025-01-03; First posted 2025-01-15 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Complications; Heart Failure
Keywords: Liver Infusion Flow; postoperative complication; transthoracic echocardiography; transesophageal echography; Swan-Ganz catheter; portal vein flow; Right Ventricular Dysfunction
MeSH Terms: conditions — Postoperative Complications; Heart Failure; Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transthoracic and Transesophageal echography within 24 hours post cardiac surgery: Measurement of portal flow velocity using transthoracic echography, as well as measurement of the superior vena cava via transesophageal echography for predicting right ventricular dysfunction.
  Interventions: Other: Transthoracic and Transesophageal echography within 24 hours post cardiac surgery

INTERVENTIONS:
Other: Transthoracic and Transesophageal echography within 24 hours post cardiac surgery — Transthoracic and Transesophageal echography within 24 hours post cardiac surgery in patients at risk for postoperative complications

SUMMARY:
Right ventricular dysfunction (RVD) after cardiac surgery is associated with ischemia and myocardial injury. While echocardiographic measures like Tricuspid Annular Plane Systolic Excursion (TAPSE) are frequently used to assess ventricular function, they have limitations in terms of accuracy. The pulmonary artery catheter remains the gold standard for assessing RVD.

This dysfunction is associated with an increased risk of both renal and hepatic failure, complications that significantly affect patient outcomes. Doppler ultrasound has emerged as a valuable tool in predicting these complications, particularly in monitoring portal circulation and hepatic perfusion.

This study aims to explore the association between portal flow pulsatility and RVD after cardiac surgery.

DETAILED DESCRIPTION:
The postoperative right ventricular dysfunction (RVD) after cardiac surgery has been described since the 1990s. It is associated to various pathophysiological mechanisms, including ischemia from prolonged aortic clamping, cardioplegia defects, myocardial injury, and ischemia-reperfusion phenomena.

Many studies have observed reduced right ventricular function intraoperatively through transthoracic echocardiographic parameters like TAPSE, fractional area change, and longitudinal strain. However, accurately assessing RVD is challenging, as these parameters can be affected post-surgery without indicating true ventricular failure.

In this context, obtaining reliable and robust invasive hemodynamic measurements is crucial for accurate assessment of RVD.

The pulmonary artery catheter (PAC), or Swan-Ganz catheter remains the gold standard, providing precise information on right ventricular systolic and diastolic function, pulmonary artery pressures, left ventricular end-diastolic pressure, venous oxygen saturation, and cardiac output.

In cardiac surgery, venous congestion resulting from right ventricular dysfunction is closely associated with increased mortality, leading to renal and hepatic failure. Tools like Doppler ultrasound (of renal, portal, and hepatic veins) can predict renal failure risk.

Researchers developed the VEXUS score in 2020 to assess this risk, and recent research found an association between 50% portal flow pulsatility and RVD.

However, some aspects remain to be clarified, such as the significant association between portal venous flow pulsatility and altered TAPSE.

This prospective study aims to examine the association between portal flow pulsatility and right ventricular dysfunction after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged at least 18 years
* Patients undergoing cardiac surgery with cardiopulmonary bypass and presenting at least one risk factor for postoperative complications, including:

  * Patient over 60 years old
  * Preoperative left ventricular ejection fraction (LVEF) < 50%
  * Surgery involving both coronary artery bypass grafting and valve procedures
  * Mitral valve surgery
  * Preoperative creatinine clearance less than 30 ml/min
* Patient having signed the informed consent form in accordance with regulations
* Patient covered by social security or an equivalent healthcare system

Exclusion Criteria:

* Patient presenting a confounding factor for altered portal flow:

  * Tricuspid regurgitation greater than grade 2
  * Known cirrhosis
* Patient with intrahepatic arteriovenous malformations
* Patient at risk for pulmonary artery catheter insertion:

  * Tricuspid valve surgery
  * Pacemaker or implantable cardioverter-defibrillator in place
* Patient with an esophageal tract abnormalities contraindicating transesophageal echocardiography (TEE)
* Pregnant or breastfeeding women
* Patient unable to understand the information provided
* Patient under guardianship, curatorship, or legal protection
* Patients deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery with cardiopulmonary bypass, presenting a risk factor for complicated postoperative management due to hemodynamic instability:
  * Patients over 60 years old
  * Preoperative left ventricular ejection fraction (LVEF) < 50%
  * Surgery involving coronary artery bypass grafting and valve surgery
  * Mitral valve surgery
  * Preoperative creatinine clearance less than 30 ml/min
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Measure of Portal Vein Flow Pulsality | First 24 hours post cardiac surgery
  Measured by pulsed Doppler and calculated by the following formula: FP = (Vmax - Vmin) / Vmax × 100.
Right ventricular (RV) function assessement | First 24 hours post cardiac surgery
  Right ventricular (RV) function will be assessed through invasive hemodynamic parameters measured by a pulmonary artery catheter.

SECONDARY OUTCOMES:
RV dysfunction | Maximum 30 days post cardiac surgery
  Will be evaluated with echocardiographic parameters:
  1. The systolic function is defined by the systolic excursion of the tricuspid annulus (TAPSE) < 17 mm and/or the systolic velocity of the tricuspid annulus (S' wave) < 9 cm/s.
  2. Diastolic function is assessed by analyzing the tricuspid flow with pulsed tissue Doppler, where the E/A ratio is < 0.8, or an E/A ratio between 0.8 and 2 associated with an E/E' ratio > 6, or an E/A ratio > 2 with a Tei index (TDE) < 120 ms.
Venous congestion | Maximum 30 days post cardiac surgery
  Venous congestion is measured via central venous catheter, or by echocardiographic findings
Renal failure | Maximum 30 days post cardiac surgery
  Acute kidney injury (AKI) will be defined according to the KDIGO classification.
Liver failure | Maximum 30 days post cardiac surgery
  As defined
  1. Hyperbilirubinemia > 2 mg/dL
  2. Elevated liver enzymes (AST > 110 U/L and ALT > 190 U/L)
Association Between Portal Flow and Postoperative Complications, Including Cardiac Tamponade | Maximum 30 days post cardiac surgery
  Evaluation of the occurrence of cardiac tamponade.
Association between Portal Flow and Postoperative complications, Including Cardiac arrhythmias | Maximum 30 days post cardiac surgery
  Evaluation of the occurrence of ventricular arrhythmias.
Association between Portal Flow and Postoperative complications, Including initiation of extracorporeal renal replacement therapy | Maximum 30 days post cardiac surgery
  Evaluation of the occurrence of the need for initiation of extracorporeal renal replacement therapy (RRT)
Association between Portal Flow and Postoperative complications, Including mechanical ventilation | Maximum 30 days post cardiac surgery
  Use of ventilatory support through mechanical ventilation
Association between Portal Flow and Postoperative complications, Including catecholamine administration | Maximum 30 days post cardiac surgery
  Evaluation of the occurrence of catecholamine administration
Association between Portal Flow and Postoperative complications, Including mortality | Maximum 30 days post cardiac surgery
  Mortality in the ICU and in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- CMC Ambroise Paré Hartmann, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No